CLINICAL TRIAL: NCT02981446
Title: A Phase III, Randomized, Observer-Masked, Active-Controlled, Parallel-Group, Multinational and Multicenter Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution 0.002% Compared With Latanoprost Ophthalmic Solution 0.005% in Subjects With Open-Angle Glaucoma or Ocular Hypertension- PEONY Study
Brief Title: A Phase III Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution Compared With Latanoprost Ophthalmic Solution in Subjects With OAG or OHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01171505
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2019-06

CONDITIONS: Open Angle Glaucoma or Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DE-117 ophthalmic solution (Experimental)
  Interventions: Drug: DE-117
- Latanoprost ophthalmic solution 0.005% (Active Comparator)
  Interventions: Drug: Latanoprost ophthalmic solution

INTERVENTIONS:
Drug: DE-117 — DE-117 ophthalmic solution will be taken one drop, once daily for 3 months in both eyes.
  Arms: DE-117 ophthalmic solution
Drug: Latanoprost ophthalmic solution — Latanoprost ophthalmic solution will be taken one drop, once daily for 3 months in both eyes.
  Other Names: Xalatan
  Arms: Latanoprost ophthalmic solution 0.005%

SUMMARY:
The purpose of this study is to investigate the intraocular pressure-lowering effect and the safety of DE-117 ophthalmic solution compared with Latanoprost ophthalmic solution in subjects with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open angle glaucoma or ocular hypertension in both eyes

Exclusion Criteria:

* Patients at risk of progression of visual field loss
* Patients with severe visual field defect
* Patients with any diseases that preclude participation in this study for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DE-117 Ophthalmic Solution | Latanoprost Ophthalmic Solution 0.005%
Started | 185 | 185
Completed | 170 | 177
Not Completed | 15 | 8

BASELINE CHARACTERISTICS:
Population: All 370 subjects received at least 1 dose of their assigned study medication and were included in the Safety population. Data for all subjects except 1 were included in the Full Analysis Set (FAS); 1 subject in the DE-117 arm was excluded from the FAS due to no data for at least 1 post-baseline IOP measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | DE-117 Ophthalmic Solution | Latanoprost Ophthalmic Solution 0.005% | Total
Number analyzed (Participants) | 184 | 185 | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 137 | 143 | 280
  >=65 years | 47 | 42 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.9) | 52.6 (13.1) | 53.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 97 | 175
  Male | 106 | 88 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 166 | 173 | 339
  Unknown or Not Reported | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 184 | 185 | 369
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 98 | 103 | 201
  South Korea | 21 | 20 | 41
  Singapore | 17 | 9 | 26
  Taiwan | 48 | 53 | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP at Month 3
Description: The IOP (mmHg) measured in the study eye (identified at Day 1 [baseline]) was the efficacy measure for this study. The IOP was measured using a calibrated Goldmann applanation tonometer preferably by the same Investigator (operator) and the same authorized study staff (recorder) during the study for each subject.
Time Frame: Month 3 (average of IOP at 3 time points: 09:00, 13:00, 17:00)
Population: One subject in the DE-117 arm was excluded from the FAS due to no data for at least 1 post-baseline IOP measurement.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 184 | 185
mmHg | 17.5 (0.25) | 16.8 (0.25)

2. Secondary Outcome: IOP at 9 Timepoints (First Key Secondary Efficacy Endpoint)
Description: as for outcome 1
Time Frame: 09:00, 13:00, and 17:00 at Week 1, Week 6, and Month 3.
Population: One subject in the DE-117 arm was excluded from the FAS due to no data for at least 1 post-baseline IOP measurement.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 184 | 185
mmHg
  Week 1 09:00: number analyzed (Participants) | 183 | 185
  Week 1 09:00 | 19.0 (0.28) | 18.8 (0.29)
  Week 1 13:00: number analyzed (Participants) | 183 | 184
  Week 1 13:00 | 18.4 (0.28) | 18.4 (0.29)
  Week 1 17:00: number analyzed (Participants) | 183 | 184
  Week 1 17:00 | 18.0 (0.28) | 18.3 (0.28)
  Week 6 09:00: number analyzed (Participants) | 176 | 180
  Week 6 09:00 | 17.8 (0.26) | 17.4 (0.26)
  Week 6 13:00: number analyzed (Participants) | 174 | 181
  Week 6 13:00 | 17.6 (0.27) | 17.2 (0.27)
  Week 6 17:00: number analyzed (Participants) | 174 | 180
  Week 6 17:00 | 17.5 (0.26) | 17.1 (0.27)
  Month 3 09:00: number analyzed (Participants) | 170 | 176
  Month 3 09:00 | 17.9 (0.27) | 17.0 (0.27)
  Month 3 13:00: number analyzed (Participants) | 170 | 176
  Month 3 13:00 | 17.2 (0.25) | 16.7 (0.26)
  Month 3 17:00: number analyzed (Participants) | 170 | 176
  Month 3 17:00 | 17.2 (0.26) | 16.7 (0.27)

3. Secondary Outcome: Mean Diurnal IOP at Week 1 (Second Key Secondary Endpoint)
Description: as for outcome 1
Time Frame: Week 1
Population: One subject in the DE-117 arm was excluded from the FAS due to no data for at least 1 post-baseline IOP measurement.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 184 | 185
mmHg | 18.5 (0.26) | 18.5 (0.27)

ADVERSE EVENTS:
Time Frame: An on-study AE were reported after the date of informed consent through the last study visit at Month 3. An AE was considered as treatment-emergent if the AE occurred on or after the treatment start date up to the last study visit. Treatment-emergent AEs were a subset of on-study AEs. AE reporting was executed until last study visit, 3 months later after randomization.
Description: Regardless of relationship to the investigational medicinal product, an AE is an unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product. Adverse events were coded using the Medical Dictionary for Regulatory Activities (MedDRA; Version 19.0).
Arm/Group | DE-117 Ophthalmic Solution | Latanoprost Ophthalmic Solution 0.005%
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/185
Serious Adverse Events (participants affected / at risk) | 2/185 | 2/185
Other Adverse Events (participants affected / at risk) | 74/185 | 55/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DE-117 Ophthalmic Solution (N=185) | Latanoprost Ophthalmic Solution 0.005% (N=185)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-117 Ophthalmic Solution (N=185) | Latanoprost Ophthalmic Solution 0.005% (N=185)
Conjunctival hyperaemia (Eye disorders) | 22 | 10
Photophobia (Eye disorders) | 10 | 1
Dry eye (Eye disorders) | 9 | 4
Corneal thickening (Eye disorders) | 7 | 2
Eye pain (Eye disorders) | 5 | 6
Ocular hyperaemia (Eye disorders) | 4 | 4
Vision blurred (Eye disorders) | 4 | 2
Conjunctival irritation (Eye disorders) | 3 | 1
Corneal deposits (Eye disorders) | 3 | 0
Eye irritation (Eye disorders) | 3 | 2
Corneal pigmentation (Eye disorders) | 2 | 0
Eye discharge (Eye disorders) | 2 | 0
Eye pruritus (Eye disorders) | 2 | 4
Eyelid irritation (Eye disorders) | 2 | 1
Eyelids pruritus (Eye disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 2 | 1
Conjunctival follicles (Eye disorders) | 1 | 0
Corneal erosion (Eye disorders) | 1 | 1
Corneal opacity (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 1
Foreign body sensation in eyes (Eye disorders) | 1 | 3
Iritis (Eye disorders) | 1 | 0
Noninfective conjunctivitis (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 2
Uveitis (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Blepharal pigmentation (Eye disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eyelash thickening (Eye disorders) | 0 | 1
Growth of eyelashes (Eye disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 3 | 5
Nasopharyngitis (Infections and infestations) | 1 | 4
Stoma site infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Optic nerve cup/disc ratio increased (Investigations) | 1 | 0
Vital dye staining cornea present (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT02981446/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02981446/SAP_001.pdf